CLINICAL TRIAL: NCT03112044
Title: Lung Transplantation Using Hepatitis C Positive Donors to Hepatitis C Negative Recipients: A Pilot Study
Brief Title: Lung Transplant HCV, Pilot Study
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-6084; UHNTID006 (Other: Tx ID research)
Record Dates: First submitted 2017-04-06; First posted 2017-04-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Lung Transplant Infection; Hepatitis C
Keywords: Lung; Transplant; Hepatitis C; DAAs; Epclusa
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Intervention Model Description: Investigators aim to transplant 20 HCV- recipients with end-stage lung disease from transplant wait-list using lungs from HCV+ donors. Donor lungs will be selected based on usual donor selection criteria evaluating blood gas analysis, chest imaging, bronchoscopy findings, and assessment in the operating room. Once lungs meet criteria for transplantation, they will be retrieved in standard fashion, transported to Toronto General Hospital in cold static preservation, placed on EVLP for 6 hours, and transplanted to consented recipients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HCV+ lung transplant to HCV- recipients (Experimental): HCV+ donor lungs will be treated with Normothermic Ex Vivo Lung Perfusion (EVLP) in order to reduce viral load and minimize risk of HCV transmission. Patients who become viremic defined as at least two consecutive positive samples will receive sofosbuvir/velpatasvir 400 mg/100 mg (Epclusa) for 12 weeks.
  Interventions: Drug: Sofosbuvir-velpatasvir (400 mg/100 mg); Device: Ex Vivo Lung Perfusion (EVLP)

INTERVENTIONS:
Drug: Sofosbuvir-velpatasvir (400 mg/100 mg) — Patients will have standard monitoring with HCV RNA and liver panel assessment at 2 week intervals until HCV is undetectable and then at the end of treatment and 3 and 6 months following its completion. Post-operative transplant care and immunosuppression will be carried on as usual transplant practice at Toronto General Hospital.
  Other Names: Epclusa
Device: Ex Vivo Lung Perfusion (EVLP) — Normothermic EVLP is a method of donor lung preservation, assessment, treatment, and repair of injured organs. This method allows donor lungs to be treated for at least 12h under protective physiological conditions.
  Other Names: Normothermic EVLP

SUMMARY:
In this study HCV negative recipients will be transplanted with HCV positive lungs. Investigators will attempt to decrease infectivity rates by performing Normothermic Ex vivo Lung Perfusion (EVLP), which is an approved method of donor lung preservation, assessment and treatment, and could be an excellent platform to reduce/eliminate hepatitis C virus. Patients will be treated by the standard approved direct-acting antivirals (DAAs) if infection occurs. It is planned to enroll 20 patients from the Lung transplant wait list in this study. Patients will be actively followed for 6 months including HCV PCR tests and then for up for 5 years to look for evidence of HCV infection and any liver or extra-hepatic complications, as well as standard post-transplant complications. This will be a single center pilot study.

DETAILED DESCRIPTION:
The success of lung transplantation (LTx) is significantly hindered by the lack of sufficient number of available donors. Many potential donor lungs cannot be utilized in clinical transplantation because donors have chronic viral infections such as hepatitis C (HCV) infection. This study will test the possibility of safely transplanting lungs from HCV positive donors. Donor lungs will be subjected to Normothermic Ex vivo Lung Perfusion (EVLP) for 6 hours for organ assessment and reduction of viral load prior to transplantation. After transplantation, recipients will be carefully monitored for HCV infection and if infection occurs, they will be promptly treated with highly effective antiviral therapy using newly approved DAAs. The aim of the study is to show that transplantation of lungs from HCV positive donors is safe in the era of DAAs. The hypothesis is that the rate of HCV transmission to recipients will be lower than previously described due to EVLP pre-treatment and any HCV transmission that does occur will be readily treatable and curable. If successful, the knowledge from this study can have a large impact to patients with end stage organ diseases by providing a large novel source of donors for lung and potentially other organ transplantations.

ELIGIBILITY:
Inclusion Criteria:

* Recipients listed for single or bilateral lung transplant
* HCV Nucleic Acid Amplification Testing (NAT) negative
* Ability to provide written informed consent

Exclusion Criteria:

* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety of transplantation from HCV positive donors to HCV negative recipients | 6 months
  Safety of transplantation using HCV positive donors reflected by 6 month survival and being free of HCV by PCR (either due to lack of transmission or as a result of treatment).

SECONDARY OUTCOMES:
Incidence of HCV transmission | 6 months
  Incidence of donor to recipient HCV transmission.
Correlation between viral loads and recipient infection | 6 months
  Correlation between donor viremia, EVLP perfusate virus load (PCR), lung tissue virus load at the end of EVLP (PCR) and recipient infection
Time to viremia development | 6 months
  Interval of time from transplantation to development of viremia
HCV cure rates | 6 months
  HCV cure rates after treatment of infected patients

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Cypel, MD MSc FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cypel M, Feld JJ, Galasso M, Pinto Ribeiro RV, Marks N, Kuczynski M, Kumar D, Bahinskaya I, Bagnato VS, Kurachi C, Slutsky AS, Yeung JC, Donahoe L, de Perrot M, Yasufuku K, Pierre A, Binnie M, Chaparro C, Martinu T, Chen M, Tikkanen J, Chow CW, Sidhu A, Waddell TK, Keshavjee S, Singer LG, Humar A. Prevention of viral transmission during lung transplantation with hepatitis C-viraemic donors: an open-label, single-centre, pilot trial. Lancet Respir Med. 2020 Feb;8(2):192-201. doi: 10.1016/S2213-2600(19)30268-1. Epub 2019 Oct 9. PMID 31606437